CLINICAL TRIAL: NCT02962089
Title: Do Branched Chain Amino Acids Counteract Protein Energy Wasting Through Gut Microbiota Changes in Hemodialysis Patients ?
Brief Title: Microbiota and Protein-energy Wasting (MIDIWA)
Acronym: MIDIWA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Genton Graf Laurence, Associate Physician at Clinical Nutrition Unit, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CER 13-239
Record Dates: First submitted 2016-08-23; First posted 2016-11-11 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Undernutrition
Keywords: Protein-energy wasting; Hemodialysis patients; Microbiota; Branched chain amino acids; Undernutrition; Malnutrition; Renal failure; Dialysis; Protein; Appetite; Body composition; Energy expenditure
MeSH Terms: conditions — Malnutrition; Renal Insufficiency | interventions — Amino Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Isocaloric isonitrogenous placebo for 4 months (7g, twice daily)
  Interventions: Dietary Supplement: Placebo
- Branched chain amino acids (BCAA) (Active Comparator): BCAA mixture for 4 months (7g, twice daily)
  Interventions: Dietary Supplement: Branched chain amino acids (BCAA)

INTERVENTIONS:
Dietary Supplement: Branched chain amino acids (BCAA)
  Arms: Branched chain amino acids (BCAA)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Oral supplementation with branched chain amino acids (BCAA) increases the levels of circulating BCAA, stimulates BCAA uptake in muscles, and decreases amino acid release from muscle, eventually promoting muscle anabolism. However, uptake of oral BCAA by muscle is not complete, pointing out that non-muscular tissues, as the splanchnic bed and gut microbiota, may play a role in BCAA metabolism.

This protocol aims at studying the impact of protein-energy wasting (PEW) and of refeeding with branched chain amino acids (BCAA), on gut barrier including gut microbiota, in chronic hemodialysis (HD) patients. The investigators speculate that:

1. HD patients with PEW have altered composition and function of gut microbiota, increased permeability of epithelial gut barrier, increased systemic inflammation but decreased fecal immunoglobulin A (IgA), and a dysbalance of plasma appetite mediators in favor of anorexigenic mediators, compared to HD patients without PEW, non dialyzed patients with chronic kidney disease and well-nourished non obese subjects,
2. BCAA supplementation of HD patients with PEW reverses these changes, thereby improving nutritional state, physical function, quality of life and resistance to infections.

DETAILED DESCRIPTION:
General description :

This protocol is multicenter (University Hospitals of Geneva (HUG), Lausanne University Hospital (CHUV), Hospital of Sion (HVS), dialysis center of the Champel clinic in Geneva and dialysis center of the Cécil clinic in Lausanne) and encompasses two parts, a cross-sectional and a longitudinal study:

1. Cross-sectional study: It is performed to differentiate the respective impact of uremia and protein-energy wasting (PEW) on gut barrier and gut microbiota. It will compare gut barrier of hemodialysis (HD) patients with PEW, with gut barrier of age-matched HD well-nourished patients, non dialyzed patients with chronic kidney disease (CKD), and healthy non obese volunteers (10 in each group). This study part is essential for interpretation of the changes occurring in the longitudinal study.
2. Longitudinal double blind randomized crossover study: HD patients with PEW (36 patients), receive, in a randomized double-blind order, either BCAA or an isocaloric isonitrogenous placebo for 4 months each, with a wash-out period of 1 month.

Randomization :

1. Cross-sectional study: No randomization will be performed. HD patients without PEW, non dialyzed patients with CKD and healthy non obese volunteers will be included if matched for gender and age with the included HD patients with PEW. Age-matching will allow a discrepancy of +/- 5 years compared to the HD patient.
2. Longitudinal study: Sequence assignment will be randomized separately in each center to ensure an equal percentage of each sequence in both centers. For this purpose, the investigators will generate 2 lists of randomization with the method of randomly permuted blocks with random block sizes of 2 and 4.

Recruitment :

Patients will be recruited among the outpatients of the Nephrology Divisions or Services of the HUG, CHUV, HVS and Champel and Cécil clinics. Healthy volunteers will be recruited among hospital staff or their relatives.

Inclusion Criteria :

1. HD patients with PEW

   * Age ≥ 18 years.
   * Maintenance HD for at least 3 months.
   * Fasting predialysis plasma albumin < 38 g/l in the absence of an known acute infection during the last 2 weeks or body weight loss > 5% of estimated dry body weight over 3 months
   * Dietary intakes (24h dietary recall) between 20-30 kcal/kg/d and < 1 g protein/kg/d on one occasion, during screening. These intakes will not include the intake of oral nutritional supplements, as intakes below 20 kcal/kg/d request artificial nutrition.
   * Absence of any systematic antibiotic treatment for an acute infection in the month preceding the inclusion.
2. HD patients without PEW

   * Patients matched for age and gender to HD patients with PEW.
   * Maintenance HD for at least 3 months.
   * Fasting predialysis plasma albumin ≥ 40 g/l, in the absence of any known acute infection during the last 2 weeks
   * Dietary intakes (24h dietary recall) > 30 kcal/kg/d and > 1.2 g protein/kg/d, once during screening.
   * Absence of any systematic antibiotic treatment for an acute infection in the month preceding the inclusion.
3. Non dialysed patients with chronic kidney disease stage 4

   * Patients matched for age and gender to HD patients with PEW.
   * Chronic kidney disease, stage 4 or 5, not requiring HD.
   * Fasting predialysis plasma albumin ≥ 40 g/l, in the absence of any known acute infection during the last 2 weeks
   * Dietary intakes (24h dietary recall) > 30 kcal/kg/d once during screening.
   * Absence of any systematic antibiotic treatment for an acute infection in the month preceding the inclusion.
4. Healthy non obese volunteers

   * Subjects matched for age and gender to HD patients with PEW.
   * Body mass index < 30 kg/m2
   * Absence of chronic disease potentially leading to wasting or cachexia.
   * Absence of plasma C-reactive protein > 50 mg/l in the last 2 weeks or known acute infection.
   * Absence of any systematic antibiotic treatment for an acute infection in the month preceding the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Maintenance hemodialysis for at least 3 months.
* Fasting predialysis plasma albumin < 38 g/l in the absence of any known acute infection during the last 2 weeks or body weight loss > 5% of estimated dry body weight over 3 months
* Dietary intakes (24h dietary recall) between 20-30 kcal/kg/d and < 1 g protein/kg/d on one occasion, during screening. These intakes will not include the intake of oral nutritional supplements, as intakes below 20 kcal/kg/d request artificial nutrition
* Absence of any systematic antibiotic treatment for an acute infection in the month preceding the inclusion

Exclusion Criteria:

* Known psychiatric or cognitive disorder, precluding protocol compliance.
* Life expectancy below 1 year.
* Inadequate dialysis (Kt/V<1.2 on 3 consecutive occasions, for HD patients only), if applicable.
* Enteral or parenteral nutrition.
* Drugs or oral nutritional supplements containing fibers since ≤ 1 month.
* Known reasons for decreased plasma albumin levels as liver failure or exudative enteropathy.
* Drugs influencing body composition, ≤ 1 month : systemic corticosteroids, anabolic drugs as insulin or testosterone, post-menopausal hormone therapy, injectable contraceptives.
* Known endocrinological disorders potentially leading to hypo- or hypermetabolism, untreated or treated since ≤ 1 month : disorders of thyroid gland, adrenal glands...
* Pregnancy and breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition by 16-S high throughput sequencing | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Gut microbiota function by 16-S high throughput sequencing | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)

SECONDARY OUTCOMES:
Epithelial gut barrier function by fasting level of plasma glucagon-like peptide-2 | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Epithelial gut barrier function by fasting level of plasma lipopolysaccharide | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Intestinal immunity by level of fecal IgA | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Systemic inflammation by fasting level of plasma interleukin 10 | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Systemic inflammation by fasting level of plama interleukin 6 | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Systemic inflammation by fasting level of plama tumor necrosis factor alpha | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma cholecystokinin | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma leptin | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma peptide YY | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma glucagon-like peptide-1 | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma neuropeptide Y | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma ghrelin | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Appetite by fasting level of plasma endocannabinoids | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Calorie and protein intakes by 3-day food diary | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Body composition by dual-energy x-rax absorptiometry (DEXA) | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Resting energy expenditure (REE) by indirect calorimetry | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Physical activity level by 7-day pedometry | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Handgrip strength by dynamometer | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Quality of life score by Short Form Health Survey (SF-36) | Changes between baseline and end of each treatment (i.e.changes between Month 0 and Month 4 and between Month 5 and Month 9)
Body composition by bioelectrical impedance analysis | Changes between baseline and end of each treatment (i.e.changes between Month 0,2, and Month 4 and between Month 5,7 and Month 9)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton, MD, Principal Investigator — University Hospital, Geneva
Locations (5):
- Switzerland (5):
  - Cécil clinic, Lausanne, Canton of Vaud
  - Lausanne University Hospital, Lausanne, Canton of Vaud
  - Hospital of Sion, Sion, Valais
  - Geneva University Hospital, Geneva
  - Champel clinic, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genton L, Pruijm M, Teta D, Bassi I, Cani PD, Gaia N, Herrmann FR, Marangon N, Mareschal J, Muccioli GG, Stoermann C, Suriano F, Wurzner-Ghajarzadeh A, Lazarevic V, Schrenzel J. Gut barrier and microbiota changes with glycine and branched-chain amino acid supplementation in chronic haemodialysis patients. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1527-1539. doi: 10.1002/jcsm.12781. Epub 2021 Sep 18. PMID 34535959
- [Derived] Genton L, Teta D, Pruijm M, Stoermann C, Marangon N, Mareschal J, Bassi I, Wurzner-Ghajarzadeh A, Lazarevic V, Cynober L, Cani PD, Herrmann FR, Schrenzel J. Glycine increases fat-free mass in malnourished haemodialysis patients: a randomized double-blind crossover trial. J Cachexia Sarcopenia Muscle. 2021 Dec;12(6):1540-1552. doi: 10.1002/jcsm.12780. Epub 2021 Sep 14. PMID 34519439